CLINICAL TRIAL: NCT03722420
Title: A Phase III, Multi-center, Open-Label, Randomized Study of the Efficacy of Radotinib Versus Imatinib in Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myeloid Leukemia Chinese Patients in Chronic Phase
Brief Title: Randomized Evaluation of Radotinib Versus Imatinib in Phase III Study for Efficacy With Chinese Patients (RERISE China)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT51CN03
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — 4-methyl-N-(3-(4-methylimidazol-1-yl)-5-trifluoromethylphenyl)-3-(4-pyrazin-2-ylpyrimidin-2-ylamino)benzamide; Imatinib Mesylate

STUDY DESIGN:
Intervention Model Description: Parallel, 2 arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radotinib 300mg (Experimental): Oral adminstration of Radotinib 300mg BID (600mg/day) for 12months
  Interventions: Drug: Radotinib
- Imatinib 400mg (Active Comparator): Oral administration of Imatinib 400mg QD (400mg/day) for 12months
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Radotinib — Patients randomized to the radotinib arms will receive 300 mg of radotinib BID (1 in the morning and 1 in the evening, at approximately 12-hour intervals).
  Other Names: Supect
  Arms: Radotinib 300mg
Drug: Imatinib — Patients randomized to the imatinib 400 mg arm will receive imatinib once a day throughout the study.
  Other Names: Glivec
  Arms: Imatinib 400mg

SUMMARY:
This is a Phase III, multi-center, open-label, parallel, 2-arm, randomized study to evaluate the efficacy and safety of radotinib 300 mg Bis In Die(BID) versus imatinib 400 mg Quaque Die(QD).

This study will be conducted in Chinese patients with newly diagnosed Ph+ Chronic Myelogenous Leukemia(CML)-Chronic Phase(CP) who are previously untreated for Chronic Myelogenous Leukemia(CML).

DETAILED DESCRIPTION:
Patients randomized to the radotinib arms will receive 300 mg of radotinib BID at approximately 12-hour intervals. Patients randomized to the imatinib 400 mg arm will receive imatinib once a day throughout the study.

The primary efficacy endpoint is the rate of Major Molecular Response(MMR) at 12 months (1 month = 4 weeks = 28 days), defined as BCR ABL1/ABL% ≤ 0.1% by international scale. The Molecular Response(MR) rate will be measured every 3 months by Real-time Quantitative(RQ)-Polymerase Chain Reaction(PCR) in a central laboratory. All patients will be treated and/or followed for 12 months (48 weeks) after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. China who are 18 years of age or older.
2. Eastern cooperative oncology group (ECOG) score 0, 1, or 2.
3. Patients with confirmed diagnosis of CML-CP within last 6 months.
4. Patients with cytogenetically confirmed Ph+ CML in chronic phase
5. Patients with typical BCR-ABL1 transcript type such as b2a2 and b3a2.
6. Patients with adequate organ function.
7. Women of childbearing potential should have negative serum or urine pregnancy test within 14 days before study entry.
8. Patients providing written informed consent before initiation of any study-related activities.

Exclusion Criteria:

1. Patients with Philadelphia chromosome negative but BCR-ABL1 positive CML.
2. Patients who had been treated with interferon or other targeted anti-cancer therapy which inhibits the growth of leukemic cells
3. Concurrently clinically significant primary malignancy
4. Patients who previously received radiotherapy
5. Patients with impaired cardiac function.
6. uncontrolled chronic medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2018-12-28 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The MMR rate | at 12 months after radotinib or imatinib treatment
  The MMR rate at 12 months after radotinib or imatinib treatment in patients with newly diagnosed CML-CP.

SECONDARY OUTCOMES:
MMR rate | by 3, 6, 9, and 12 months of treatment.
  To compare MMR rate for the best response in patients within specific periods.
Complete Cytogenetic Response(CCyR) rate | by 3, 6, 9, and 12 months of treatment.
  To compare CCyR rate for the best response in patients within specific periods.
The MR 4.0 and MR 4.5 rates | by 3, 6, 9, and 12 months of treatment, and late
  To compare the MR4.0 and MR4.5 rates for the best response in patients within specific periods.
Disease progression (AP/BC) rate | at 3, 6, and 12 months
  To compare disease progression for the best response in patients within specific periods.
Failure rate according to European Leukemia Net (ELN) guideline 2013 (ELN 2013*) | at 3, 6, and 12 months
  To compare failure rate for the best response in patients within specific periods.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Qian, Principal Investigator — Peking University People's Hospital(北京大学人民医院)
Locations (1):
- Peking University People's Hospital(北京大学人民医院), Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided